CLINICAL TRIAL: NCT01610739
Title: Effect of Carpal Tunnel Release on Median Nerve Perfusion Using SPY Scope Imaging
Brief Title: Carpal Tunnel Release Effects on Median Nerve Perfusion
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: never initiated; did not recruit patients
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Nadia M. Obeid, MD, M.D., Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HFHSobeid2012
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Median nerve perfusion (Other): Injection of indigocyanine green dye to evaluate perfusion of the median nerve with the SPY scope before and after carpal tunnel release
  Interventions: Drug: Indigocyanine green dye

INTERVENTIONS:
Drug: Indigocyanine green dye — Each patient will receive 1 injection of indigocyanine green dye using 2.5 mg/mL concentration of the imaging agent. 3mL of this mixture will be injected intravenously, followed by 10mL NS bolus, just prior to imaging with the SPY scope
  Other Names: Indigocyanine green dye (ICG)

SUMMARY:
This study aims to examine the effect of carpal tunnel release on blood flow to the median nerve using SPY scope imaging to view the perfusion to the nerve.

DETAILED DESCRIPTION:
The study will involve patients undergoing carpal tunnel release surgery at our institution, with no change in the actual procedure performed. Using the SPY Scope, we will measure blood flow prior to the carpal tunnel release, and again measure once carpal tunnel release has been performed, in order to compare the values. This may add roughly 15 minutes to the total procedure time, however, no steps in the actual operation will be altered or affected in any way.

ELIGIBILITY:
Inclusion Criteria:

* carpal tunnel syndrome
* 18 years or older

Exclusion Criteria:

* pregnant
* less than 18 years of age
* allergy to iodide or iodinated contrast agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Effect of median nerve perfusion with carpal tunnel release | intraoperatively
  This study aims to examine the effect of carpal tunnel release on blood flow to the median nerve using SPY scope imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia M Obeid, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States